CLINICAL TRIAL: NCT05633017
Title: Measuring Exercise Performance and Perception With Facemask Resistance
Brief Title: Breathing With a Facemask Exercise Performance
Status: Completed | Type: Observational
Sponsor: CereVu Medical, Inc. (Industry)
Collaborators: John Muir Health (Other)
Responsible Party: Sponsor
Other Study IDs: CIP5002
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pulmonary Rehab Patients: Patients who attend respiratory therapy at John Muir Pulmonary Rehab facility
  Interventions: Combination Product: CereVu Objective Dyspnea Score
- Control: Healthy adults, 18+
  Interventions: Combination Product: CereVu Objective Dyspnea Score

INTERVENTIONS:
Combination Product: CereVu Objective Dyspnea Score — Small forehead wearable and mobile app

SUMMARY:
This study will determine the dyspnea response in chronic lung disease volunteers during treadmill walking with and without added inspiratory resistance. This study will also determine the level of dyspnea and exercise sense of effort in individuals walking on a treadmill when elevations occur. Comparisons will be made of a participant's exercise response with and without increased inspiratory resistance. In this study, exercise performance will be analyzed based on physiological and perceptual measures. The participant will undergo two sessions: one session will be a standard exercise walking test without an inspiratory resistance; the other session will be the same standard exercise walking test while breathing with an inspiratory resistance equal to a N95 facemask (R=10-15 cmH2O/L/sec). Performance will be determined by physiological measures. Perception will be determined by scores based on numerical scales and automatically with the forehead Vitality remote monitoring sensor.

ELIGIBILITY:
Inclusion Criteria:

* Former pulmonary rehabilitation patients that are now participating in maintenance exercise classes
* Males and females with an age range of 18 years or older
* Subjects must be able to walk on treadmill for multiple sessions

Exclusion Criteria:

* The subjects in each experiment will be recruited for a distribution of gender, ethnicity and age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing respiratory therapy at John Muir Health which encompasses a variety of pulmonary conditions
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-12-17 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
Correlation between dyspnea as measured by the device and reported dyspnea by subjects | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Akhbardeh, PhD, Study Director — CereVu Medical
Locations (1):
- John Muir Health, Pleasant Hill, California, United States

IPD SHARING:
Plan to Share IPD: No